CLINICAL TRIAL: NCT01726660
Title: Pilot Study of the Effects of Protocol-Specific Robotic Arm Therapy in Stroke Recovery
Brief Title: The General Use of Robots in Stroke Recovery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unfunded
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Bruce Volpe, Principal Investigator, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-121B
Record Dates: First submitted 2012-10-26; First posted 2012-11-15 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Stroke
Keywords: Stroke; Cerebrovascular Accident; Cerebral stroke; CVA; robotic therapy; upper extremity recovery; kinematic training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- IMT Robotic Arm Therapy: Aim training (Experimental): Alternating sessions of planar (shoulder/elbow) and wrist robotic therapy programmed for aim training, 3x/week for 12 weeks.
  Interventions: Device: IMT Robotic Arm therapy
- IMT Robotic Arm Therapy: Smoothness Training (Experimental): Alternating sessions of planar (shoulder/elbow) and wrist robotic therapy programmed for smoothness training, 3x/week for 12 weeks.
  Interventions: Device: IMT Robotic Arm therapy
- IMT Robotic Arm Therapy: Impairment training (Experimental): Alternating sessions of planar (shoulder/elbow) and wrist robotic therapy programmed for whole-arm, impairment training, 3x/week for 12 weeks.
  Interventions: Device: IMT Robotic Arm therapy
- IMT Robotic Arm Therapy: Functional training (Experimental): Alternating sessions of planar (shoulder/elbow) and wrist robotic therapy programmed for whole arm, functional training, 3x/week for 12 weeks.
  Interventions: Device: IMT Robotic Arm therapy

INTERVENTIONS:
Device: IMT Robotic Arm therapy — Interactive Motion Technologies (IMT) planar and wrist robots for robotic arm therapy

SUMMARY:
The purpose of this study is to determine if tailoring multiple sessions of upper extremity robotic therapy to focus on a particular aspect of movement (e.g smoothness vs. aiming; active range of motion vs. functional practice)can optimize therapeutic results and lead to greater functional returns in arm mobility after stroke.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* First single focal unilateral lesion with diagnosis verified by brain imaging, which occurred at least 6 months prior
* Cognitive function sufficient enough to understand experiments and follow instructions
* Fugl Meyer assessment at admission of 7 to 38 out of 66 (neither hemiplegic nor fully recovered motor function in the muscles of the shoulder, elbow, and wrist)

Exclusion Criteria:

* Prior experience with robotic arm therapy
* Fixed contraction of the affected limb
* Complete flaccid paralysis of the affected limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Upper Extremity Fugl Meyer Motor Assessment | 12 weeks (immediately following the intervention) and 24 weeks (3 months after the intervention)

SECONDARY OUTCOMES:
Change from baseline in Kinematic Data | 12 weeks (immediately following the intervention) and 24 weeks (3 months after the intervention)
  Kinematic Data recorded during therapy with IMT robots
Change from baseline in Fugl Meyer Sensation Scale | 12 weeks (immediately following the intervention) and 24 weeks (3 months after the intervention)
Change from baseline in Fugl Meyer Proprioception Scale | 12 weeks (immediately following the intervention) and 24 weeks (3 months after the intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce T Volpe, MD, Principal Investigator — Feinstein Institute for Medical Research
Locations (1):
- Feinstein Institute for Medical Research, Manhasset, New York, United States

REFERENCES:
- [Background] Stein J, Krebs HI, Frontera WR, Fasoli SE, Hughes R, Hogan N. Comparison of two techniques of robot-aided upper limb exercise training after stroke. Am J Phys Med Rehabil. 2004 Sep;83(9):720-8. doi: 10.1097/01.phm.0000137313.14480.ce. PMID 15314537